CLINICAL TRIAL: NCT01530815
Title: Intraoperative Local Anesthesia for Management of Postoperative Pain Following Laparoscopic Ventral Hernia Repair: a Prospective Double-blind Randomized Trial
Brief Title: Bupivicaine to Reduce Postoperative Pain in Laparoscopic Ventral Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang, Steve S., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LapHernia_SBCH
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bupivicaine Infusion (Experimental): We will infuse bupivicaine between the abdominal wall and mesh to try and reduce postoperative pain
  Interventions: Drug: Bupivicaine Infusion

INTERVENTIONS:
Drug: Bupivicaine Infusion — Investigators and Caregivers will be blinded to either 0.9% Normal Saline or 0.5% Bupivicaine infusion between the mesh and abdominal wall
  Other Names: Marcaine

SUMMARY:
The investigators are testing to see if infusion of bupivicaine between the mesh and abdominal wall can reduce postoperative pain and decrease use of narcotics in the postoperative setting.

DETAILED DESCRIPTION:
The primary objective of this study is to test different methods for pain management following laparoscopic ventral hernia repair. We hypothesize that local analgesic injection between the abdominal wall and mesh intraoperatively during laparoscopic ventral hernia repair will result in a 20% decrease in the use of post-surgery pain medication in the first four hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be scheduled for a laparoscopic ventral hernia repair at SBCH. If any additional procedure is performed, the subject will be excluded from the study
2. Age 18 or older
3. Patient must agree to complete pain journal postoperatively
4. Informed consent signed and dated by patient. Consenting through a legally authorized guardian will not be accepted due to the necessity of completing a subjective pain journal

Exclusion Criteria:

1. Any surgical procedure occurring besides the study procedure
2. Any allergy or sensitivity to bupivicaine or its derivatives
3. Less than 18 years of age
4. Patient unable to self report in pain journal due to cognitive disabilities
5. Discharged less than 4 hours post-surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hours
  We will measure pain based on pain journal and usage of postoperative pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Steve S Chang, MD, Principal Investigator — Santa Barbara Cottage Hospital
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States

REFERENCES:
- [Derived] Gough AE, Chang S, Reddy S, Ferrigno L, Zerey M, Grotts J, Yim S, Thoman DS. Periprosthetic Anesthetic for Postoperative Pain After Laparoscopic Ventral Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2015 Sep;150(9):835-40. doi: 10.1001/jamasurg.2015.1530. PMID 26154700